CLINICAL TRIAL: NCT03859284
Title: Clinical Evaluation of a Moist Bonding Self-Adhering Flowable Composite With and Without Adhesive System Versus Conventional Flowable Composite in Cervical Caries Lesions: Randomized Clinical Trial
Brief Title: Evaluation of Adhering Flowable Composite With and Without Adhesive Vs Flowable in Cervical Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mounir Ibrahim Hassan, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mon15
Record Dates: First submitted 2019-02-12; First posted 2019-03-01 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Dental Restoration Failure
MeSH Terms: interventions — Adhesives

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- flowable resin-composite (Active Comparator): 3M flowable composite is a conventional restoration to treat anterior carious cervical lesions. considered to be the gold standard of the flowable composites.
  other names: ''flowable composite ''
  Interventions: Other: flowable resin composite
- self-adhering flowable (Experimental): intervention one is moist bonding self adhering flowable composite that binds to tooth without an adhesive system
  Interventions: Other: self adhering flowable
- self-adhering flowable with adhesive (Experimental): intervention two moist bonding self adhering flowable composite that binds to tooth with the aid of adhesive system to improve the clinical performance
  Interventions: Other: self adhering flowable with adhesive

INTERVENTIONS:
Other: flowable resin composite — gold standard
  Other Names: conventional flowable composite
  Arms: flowable resin-composite
Other: self adhering flowable — moist bonding self adhering flowable composite
  Other Names: embrace wet bond
  Arms: self-adhering flowable
Other: self adhering flowable with adhesive — moist bonding self adhering flowable composite with the aid of an adhesive system.
  Other Names: embrace wet bond with adhesive
  Arms: self-adhering flowable with adhesive

SUMMARY:
With limited evidence-based information in literature about using self-adhering flowable composite in conservative class V restorations, it was found beneficial to evaluate the newly introduced material using a randomized controlled clinical trial to test the null hypothesis that moist bonding self-adhering flowable composite with and without adhesive system will have the same clinical performance as conventional flowable composite in cervical caries lesions.

DETAILED DESCRIPTION:
flowable composite is considered a gold standard in class V restorations due to its resilient character the prevents its dislodgement in this area. self-adhering flowable composite would simplify the clinical steps and claims to improve the adhesion.

ELIGIBILITY:
Inclusion Criteria:

* patients with anterior cervical carious lesions.
* Pulp asymptomatic vital carious anterior teeth.
* Co-operative patients approving to participate in the trial.

Exclusion Criteria:

* Pregnancy.
* Disabilities.
* Systemic disease or severe medical complications.
* Deep extensive carious cavities that may lead to the fracture of the tooth or pulpal affection.
* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.
* Heavy smokers.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the clinical performance using Fédération Dentaire Internationale' (FDI) World Dental Federation clinical criteria for the evaluation of the direct restoration. (FDI) criteria includes | Change from the baseline at 6 months and12 months]
  Biological properties (Postoperative hypersensitivity & tooth vitality, Recurrence of caries, erosion & abfraction,Tooth integrity (enamel cracks or tooth fractures),Periodontal response (compared to a reference tooth),Adjacent mucosa, Oral & general health).
  Esthetic properties (Surface luster, Staining (surface &margin),Color match & translucency & Esthetic anatomical form).
  Functional properties (Fracture or material retention, Marginal integrity, Occlusal contour &wear (quantitatively & qualitatively), Proximal anatomical form(contact point &contour), Radiographic examination(when applicable) &Patient's view
  For each criteria one score will be chosen from 5 scores (excellent, good, satisfactory, unsatisfactory & poor).
  Subscales will not be combined

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Giza, Egypt